CLINICAL TRIAL: NCT00570063
Title: A Phase 2, Multicenter, Double-blind, Randomized, Fixed Dose, Parallel Group, 3-week Inpatient Treatment Study To Evaluate The Safety, Efficacy And Pharmacokinetics Of Pf-02545920 Compared With Placebo In The Treatment Of Acute Exacerbation Of Schizophrenia
Brief Title: Double Blind, Randomized, 3 Week Inpatient Study To Evaluate The Safety & Efficacy Of PF-02545920 Compared With Placebo
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A8241006
Record Dates: First submitted 2007-12-06; First posted 2007-12-10 (Estimated); Results first posted 2017-12-20 (Actual); Last update posted 2017-12-20 (Actual); Status verified 2017-11

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; acute exacerbation; and PF-02545920
MeSH Terms: conditions — Schizophrenia | interventions — 2-((4-(1-methyl-4-pyridin-4-yl-1H-pyrazol-3-yl)phenoxy)methyl)quinoline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): PF-02545920 15 mg tablets taken twice a day by mouth for 21 days
  Interventions: Drug: PF-02545920
- 2 (Placebo Comparator): Matching placebo tablets taken twice a day by mouth for 21 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-02545920 — Participants are assigned to 15 mg oral tablets twice a day of PF-02545920 or placebo in parallel for the duration of the study which is 21 days
  Arms: 1
Drug: Placebo — Participants are assigned to 15 mg oral tablets twice a day of PF-02545920 or placebo in parallel for the duration of the study which is 21 days.
  Arms: 2

SUMMARY:
To assess the efficacy and safety of an investigational compound PF-02545920 for the treatment of schizophrenia. PF-02545920 will be more effective than placebo in reducing symptoms associated with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

1. Have a current diagnosis of schizophrenia.
2. Increase in symptoms over the past 2-4 weeks.
3. Willing to remain inpatients for the duration of the trial.

Exclusion Criteria:

1. Evidence or history of clinically significant medical problems.
2. Females of childbearing potential.
3. A primary psychiatric diagnosis other than schizophrenia.
4. A diagnosis of substance abuse or dependence in the last 6 months.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-11 (Actual); Primary Completion 2008-02-18 (Actual); Study Completion 2008-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- United States (10):
  - California Clinical Trials Medical Group, Inc., Glendale, California
  - Glendale Adventist Medical Center, Glendale, California
  - Telecare-Cresta Loma, Lemon Grove, California
  - California Clinical Trials Medical Group, Paramount, California
  - LaPaz Geropsychiatric Center, Paramount, California
  - California Clinical Trials Medical Group, San Diego, California
  - Connecticut Mental Health Center-Yale University, Clinical Neuroscience Research Unit, New Haven, Connecticut
  - CRI Worldwide, LLC, Willingboro, New Jersey
  - St. Anthony Hospital, Oklahoma City, Oklahoma
  - IPS Research Company, Oklahoma City, Oklahoma

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8241006&StudyName=Double%20Blind%2C%20Randomized%2C%203%20Week%20Inpatient%20Study%20To%20Evaluate%20The%20Safety%20%26%20Efficacy%20Of%20PF-02545920%20Compared%20With%20Placebo

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-02545920 15 Milligram (mg): Participants received single dose of PF-02545920 15 mg tablet, orally twice daily (approximately 12 hours apart) from Day 1 to Day 21 and were followed up to Day 31.
- Placebo: Participants received single dose of placebo tablet matched to PF-02545920, orally twice daily (approximately 12 hours apart) from Day 1 to Day 21 and were followed up to Day 31.
Period: Overall Study
Arm/Group | PF-02545920 15 Milligram (mg) | Placebo
Started | 24 | 11
Completed | 9 | 3
Not Completed | 15 | 8
Not completed — Adverse Event | 4 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Sponsor's Decision | 7 | 3

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all participants who were randomized to a treatment sequence and received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-02545920 15 Milligram (mg) | Placebo | Total
Number analyzed (Participants) | 24 | 11 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (9.3) | 43.1 (10.8) | 42.6 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 22 | 9 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) at Day 21: Total Score
Description: PANSS is a clinician-rated instrument for assessing the positive symptoms, negative symptoms, and general psychopathology specifically associated with schizophrenia. The scale consists of 30 items. Each item is rated on a scale from 1 (symptom not present) to 7 (symptoms extremely severe). PANSS total score is the sum of the 30 items and ranges from 30 to 210; where higher score indicates greater severity of symptoms.
Time Frame: Baseline (Day 1), Day 21
Population: Pharmacodynamic data (PD) analysis set included all participants with at least 1 dose of study medication and had a baseline value and at least 1 post dose PD measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-02545920 15 Milligram (mg) | Placebo
Number analyzed (Participants) | 24 | 11
units on a scale
  Baseline: number analyzed (Participants) | 24 | 10
  Baseline | 98.13 (12.28) | 96.10 (4.61)
  Change at Day 21: number analyzed (Participants) | 11 | 4
  Change at Day 21 | -19.82 (19.06) | -18.25 (24.09)
Statistical Analysis 1: Comparison: PF-02545920 15 Milligram (mg) vs Placebo; P-value and 90 percent confidence interval (CI) were obtained from mixed effects repeated measures analysis using covariance structures spatial power covariance structure (SP[POW]) with participant as random effect, treatment, visit, and visit-by-treatment interaction as fixed effects and baseline score as a covariate; Test type: Superiority or Other; p = 0.86, Mixed Models Analysis; Least square (LS) mean difference = -1.61, 90% CI 2-sided [-16.49 to 13.27], Standard Error of Mean 8.94

2. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) at Day 21: Positive Subscale Score
Description: PANSS is a clinician-rated instrument for assessing the positive symptoms, negative symptoms, and general psychopathology specifically associated with schizophrenia. PANSS positive subscale assesses the positive symptoms associated with schizophrenia as delusions, conceptual disorganization, and hallucinatory behavior. It consists of 7 items and each item is rated on a scale from 1 (symptoms not present) to 7 (symptoms extremely severe). PANSS positive subscale is the sum of 7 items and ranges from 7 to 49; where higher score indicates greater severity of symptoms.
Time Frame: Baseline (Day 1), Day 21
Population: PD analysis set included all participants with at least 1 dose of study medication and had a baseline value and at least 1 post dose PD measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-02545920 15 Milligram (mg) | Placebo
Number analyzed (Participants) | 24 | 11
units on a scale
  Baseline: number analyzed (Participants) | 24 | 10
  Baseline | 26.13 (3.31) | 26.50 (2.17)
  Change at Day 21: number analyzed (Participants) | 11 | 4
  Change at Day 21 | -5.55 (4.87) | -4.50 (7.55)
Statistical Analysis 1: Comparison: PF-02545920 15 Milligram (mg) vs Placebo; P-value and 90 percent CI were obtained from mixed effects repeated measures analysis using covariance structures (SP[POW]) with participant as random effect, treatment, visit, and visit-by-treatment interaction as fixed effects and baseline score as a covariate; Test type: Superiority or Other; p = 0.65, Mixed Models Analysis; LS mean difference = -1.23, 90% CI 2-sided [-5.71 to 3.24], Standard Error of Mean 2.69

3. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) at Day 21: Negative Subscale Score
Description: PANSS is a clinician-rated instrument for assessing the positive symptoms, negative symptoms, and general psychopathology specifically associated with schizophrenia. PANSS negative subscale assesses negative symptoms associated with schizophrenia as blunted affect, emotional withdrawal, poor rapport, and passive/apathetic social withdrawal. It consists of 7 items and each item is rated on a scale from 1 (symptoms not present) to 7 (symptoms extremely severe). PANSS negative subscale score is the sum of 7 items and ranges from 7 to 49, where higher score indicates greater severity of symptoms.
Time Frame: Baseline (Day 1), Day 21
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-02545920 15 Milligram (mg) | Placebo
Number analyzed (Participants) | 24 | 10
units on a scale
  Baseline | 24.17 (5.31) | 20.90 (3.54)
  Change at Day 21: number analyzed (Participants) | 11 | 4
  Change at Day 21 | -5.91 (5.86) | -4.50 (7.85)
Statistical Analysis 1: Comparison: PF-02545920 15 Milligram (mg) vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.93, Mixed Models Analysis; LS mean difference = -0.24, 90% CI 2-sided [-4.59 to 4.10], Standard Error of Mean 2.61

4. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) at Day 21: General Psychopathology Subscale Score
Description: PANSS is a clinician-rated instrument for assessing the positive symptoms, negative symptoms, and general psychopathology specifically associated with schizophrenia. PANSS general psychopathology subscale score assesses general psychopathology symptoms associated with schizophrenia as somatic concern, anxiety, guilt feelings, tension, mannerisms/posturing, depression, motor retardation, uncooperativeness, unusual thought content, disoriented, poor attention, lack of judgment/insight, disturbance of volition, poor impulse control, preoccupation, and active social avoidance. It consists of 16 items and each item is rated on a scale from 1 (symptoms absent) to 7 (extreme psychopathology). PANSS general psychopathology subscale score is the sum of 16 items and ranges from 16 to 112; where higher scores indicates greater severity of symptoms.
Time Frame: Baseline (Day 1), Day 21
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-02545920 15 Milligram (mg) | Placebo
Number analyzed (Participants) | 24 | 11
units on a scale
  Baseline: number analyzed (Participants) | 24 | 10
  Baseline | 47.83 (6.88) | 48.70 (3.59)
  Change at Day 21: number analyzed (Participants) | 11 | 4
  Change at Day 21 | -8.36 (10.04) | -9.25 (9.78)
Statistical Analysis 1: Comparison: PF-02545920 15 Milligram (mg) vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.86, Mixed Models Analysis; LS mean difference = 0.74, 90% CI 2-sided [-6.21 to 7.69], Standard Error of Mean 4.18

5. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) at Day 21: Positive Marder Factor Score
Description: PANSS subscales based on Marder factors assess negative symptoms, positive symptoms, disorganized thoughts factor, uncontrolled hostility/excitement factor, and anxiety/depression factor associated with schizophrenia. PANSS positive Marder factor score consists of 8 items and each item is rated on a scale from 1 (symptoms not present) to 7 (symptoms extremely severe). PANSS positive Marder factor score is the sum of 8 items and ranges from 8 to 56; where higher score indicating greater severity of symptoms.
Time Frame: Baseline (Day 1), Day 21
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-02545920 15 Milligram (mg) | Placebo
Number analyzed (Participants) | 24 | 11
units on a scale
  Baseline: number analyzed (Participants) | 24 | 10
  Baseline | 30.04 (3.47) | 29.20 (2.35)
  Change at Day 21: number analyzed (Participants) | 11 | 4
  Change at Day 21 | -6.18 (5.67) | -3.50 (9.15)
Statistical Analysis 1: Comparison: PF-02545920 15 Milligram (mg) vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.43, Mixed Models Analysis; LS mean difference = -2.57, 90% CI 2-sided [-7.92 to 2.79], Standard Error of Mean 3.22

6. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) at Day 21: Negative Marder Factor Score
Description: PANSS subscales based on Marder factors assess negative symptoms, positive symptoms, disorganized thoughts factor, uncontrolled hostility/excitement factor, and anxiety/depression factor associated with schizophrenia. PANSS negative Marder factor score consists of 7 items and each item is rated on a scale from 1 (symptoms not present) to 7 (symptoms extremely severe). PANSS negative Marder factor score is the sum of 7 items and ranges from 7 to 49; where higher score indicating greater severity of symptoms.
Time Frame: Baseline (Day 1), Day 21
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-02545920 15 Milligram (mg) | Placebo
Number analyzed (Participants) | 24 | 11
units on a scale
  Baseline: number analyzed (Participants) | 24 | 10
  Baseline | 22.63 (5.50) | 20.30 (4.11)
  Change at Day 21: number analyzed (Participants) | 11 | 4
  Change at Day 21 | -6.27 (5.83) | -5.75 (8.30)
Statistical Analysis 1: Comparison: PF-02545920 15 Milligram (mg) vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.91, Mixed Models Analysis; LS mean difference = -0.30, 90% CI 2-sided [-4.76 to 4.16], Standard Error of Mean 2.68

7. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) at Day 21: Disorganized Thought Marder Factor Score
Description: PANSS subscales based on Marder factors assess negative symptoms, positive symptoms, disorganized thoughts factor, uncontrolled hostility/excitement factor, and anxiety/depression factor associated with schizophrenia. PANSS disorganized thought Marder factor score consists of 7 items and each item is rated on a scale from 1 (symptoms not present) to 7 (symptoms extremely severe). PANSS disorganized thought Marder factor score is the sum of 7 items and ranges from 7 to 49; where higher score indicating greater severity of symptoms.
Time Frame: Baseline (Day 1), Day 21
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-02545920 15 Milligram (mg) | Placebo
Number analyzed (Participants) | 24 | 11
units on a scale
  Baseline: number analyzed (Participants) | 24 | 10
  Baseline | 22.92 (5.42) | 21.50 (3.41)
  Change at Day 21: number analyzed (Participants) | 11 | 4
  Change at Day 21 | -4.18 (5.10) | -3.50 (4.80)
Statistical Analysis 1: Comparison: PF-02545920 15 Milligram (mg) vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.78, Mixed Models Analysis; LS mean difference = 0.63, 90% CI 2-sided [-3.17 to 4.43], Standard Error of Mean 2.29

8. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) at Day 21: Hostility/Excitement Marder Factor Score
Description: PANSS subscales based on Marder factors assess negative symptoms, positive symptoms, disorganized thoughts factor, uncontrolled hostility/excitement factor, and anxiety/depression factor associated with schizophrenia. PANSS hostility/excitement Marder factor score consists of 4 items and each item is rated on a scale from 1 (symptoms not present) to 7 (symptoms extremely severe). PANSS hostility/excitement Marder factor score is the sum of 4 items and ranges from 4 to 28; where higher score indicating greater severity of symptoms.
Time Frame: Baseline (Day 1), Day 21
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-02545920 15 Milligram (mg) | Placebo
Number analyzed (Participants) | 24 | 11
units on a scale
  Baseline: number analyzed (Participants) | 24 | 10
  Baseline | 9.33 (3.58) | 10.80 (3.05)
  Change at Day 21: number analyzed (Participants) | 11 | 4
  Change at Day 21 | -0.45 (3.11) | -1.25 (2.06)
Statistical Analysis 1: Comparison: PF-02545920 15 Milligram (mg) vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.92, Mixed Models Analysis; LS mean difference = 0.14, 90% CI 2-sided [-2.11 to 2.39], Standard Error of Mean 1.35

9. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) at Day 21: Anxiety/Depression Marder Factor Score
Description: PANSS subscales based on Marder factors assess negative symptoms, positive symptoms, disorganized thoughts factor, uncontrolled hostility/excitement factor, and anxiety/depression factor associated with schizophrenia. PANSS anxiety/depression Marder factor score consists of 4 items and each item is rated on a scale from 1 (symptoms not present) to 7 (symptoms extremely severe). PANSS anxiety/depression Marder factor score is the sum of 4 items and ranges from 4 to 28; where higher score indicating greater severity of symptoms.
Time Frame: Baseline (Day 1), Day 21
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-02545920 15 Milligram (mg) | Placebo
Number analyzed (Participants) | 24 | 11
units on a scale
  Baseline: number analyzed (Participants) | 24 | 10
  Baseline | 13.21 (2.34) | 14.30 (2.75)
  Change at Day 21: number analyzed (Participants) | 11 | 4
  Change at Day 21 | -2.73 (3.64) | -4.25 (2.87)
Statistical Analysis 1: Comparison: PF-02545920 15 Milligram (mg) vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.60, Mixed Models Analysis; LS mean difference = 0.84, 90% CI 2-sided [-1.85 to 3.54], Standard Error of Mean 1.62

10. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) at Day 21: Derived Brief Psychiatric Rating Scale (BPRS) Core Psychosis Total Score
Description: BPRS is a clinician-rated instrument for assessing conceptual disorganization, hallucinatory behavior, suspiciousness and unusual thought content associated with schizophrenia. The scale consists of 18 items. Each item is rated on a scale from 0 (symptom not present) to 6 (symptoms extremely severe). BPRS core psychosis total score is the sum of 18 items and ranges from 0 to 108; where higher score indicates greater severity of symptoms.
Time Frame: Baseline (Day 1), Day 21
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-02545920 15 Milligram (mg) | Placebo
Number analyzed (Participants) | 24 | 11
units on a scale
  Baseline: number analyzed (Participants) | 24 | 10
  Baseline | 17.17 (2.35) | 17.60 (1.65)
  Change at Day 21: number analyzed (Participants) | 11 | 4
  Change at Day 21 | -3.55 (3.24) | -4.25 (5.50)
Statistical Analysis 1: Comparison: PF-02545920 15 Milligram (mg) vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.81, Mixed Models Analysis; LS mean difference = 0.44, 90% CI 2-sided [-2.65 to 3.53], Standard Error of Mean 1.86

11. Secondary Outcome: Change From Baseline in Clinical Global Impression Severity Scale (CGI-S) Score at Day 21
Description: CGI-S is a 7-point clinician-rated scale for assessing the global severity of schizophrenia. Score range: 1 (normal - not ill at all) to 7 (most extreme illness). Higher score indicating greater degree of illness.
Time Frame: Baseline (Day 1), Day 21
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-02545920 15 Milligram (mg) | Placebo
Number analyzed (Participants) | 24 | 11
units on a scale
  Baseline: number analyzed (Participants) | 24 | 10
  Baseline | 4.88 (0.448) | 4.9 (0.568)
  Change at Day 21: number analyzed (Participants) | 11 | 4
  Change at Day 21 | -0.91 (0.701) | -1 (1.414)
Statistical Analysis 1: Comparison: PF-02545920 15 Milligram (mg) vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.93, Mixed Models Analysis; LS mean difference = -0.04, 90% CI 2-sided [-0.84 to 0.76], Standard Error of Mean 0.48

12. Secondary Outcome: Change From Baseline in Clinical Global Impression Improvement Scale (CGI-I) Score at Day 21
Description: CGI-improvement is a 7-point clinician-rated scale for assessing the global improvement of schizophrenia ranging from 1 (very much improved) to 7 (very much worse). Higher score indicating less improvement.
Time Frame: Baseline (Day 4), Day 21
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-02545920 15 Milligram (mg) | Placebo
Number analyzed (Participants) | 24 | 11
units on a scale
  Baseline: number analyzed (Participants) | 23 | 10
  Baseline | 3.3 (0.93) | 3.6 (0.52)
  Change at Day 21: number analyzed (Participants) | 11 | 4
  Change at Day 21 | 3.09 (1.51) | 3 (1.83)
Statistical Analysis 1: Comparison: PF-02545920 15 Milligram (mg) vs Placebo; P-value and 90 percent CI were obtained from mixed effects repeated measures analysis using covariance structures (SP[POW]) with participant as random effect, treatment, visit, and visit-by-treatment interaction as fixed effects; Test type: Superiority or Other; p = 0.99, Mixed Models Analysis; LS mean difference = 0.01, 90% CI 2-sided [-1.13 to 1.14], Standard Error of Mean 0.68

13. Secondary Outcome: Change From Baseline in Nurses' Observation Scale for Inpatient Evaluation (NOSIE-30) Subscale Scores at Day 21
Description: NOSIE is an inpatient treatment staff-administered questionnaire. It consists of 30 items: 26 items divided into 6 subscales and 4 individual items. Each item is rated on a 5-point scale (0= never to 4= always), to assess functional ability of participants. 6 subscales: irritability (sum of 5 items: score range 0 to 20), manifest psychosis (sum of 4 items: score range 0 to 16), personal neatness (sum of 4 items: score range 0 to 16), retardation (sum of 3 items: score range 0 to 12), social competence (sum of 5 items: score range 0 to 20) and social interest (sum of 5 items: score range 0 to 20) and 4 individual items: cried (score range 0 to 4), refused to speak (score range 0 to 4), said felt blue or depressed (score range 0 to 4) and said he/she was no good (score range 0 to 4). For each of the 6 subscales and 4 individual items: higher scores indicates irregular functional ability.
Time Frame: Baseline (Day 1), Day 21
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-02545920 15 Milligram (mg) | Placebo
Number analyzed (Participants) | 19 | 9
units on a scale
  Baseline: Cried | 0.26 (0.933) | 0.22 (0.441)
  Change at Day 21: Cried | -0.16 (0.958) | 0 (0.5)
  Baseline: Felt blue or depressed | 0.63 (0.761) | 1.11 (1.269)
  Change at Day 21: Felt blue or depressed | 0 (0.882) | -0.44 (1.424)
  Baseline: Irritability | 2.47 (2.611) | 3.67 (5.958)
  Change at Day 21: Irritability | 1.21 (4.063) | -0.33 (4.848)
  Baseline: Manifest psychosis | 2.37 (2.314) | 3.78 (3.27)
  Change at Day 21: Manifest psychosis | -0.32 (2.868) | -0.89 (3.14)
  Baseline: Personal neatness | 11.95 (3.535) | 11.11 (4.256)
  Change at Day 21: Personal neatness | 0 (2.236) | -0.56 (1.74)
  Baseline: Refused to speak | 0.32 (0.582) | 0 (0)
  Change at Day 21: Refused to speak | -0.11 (0.567) | 0.22 (0.441)
  Baseline: Retardation | 4.05 (2.527) | 3.67 (1.323)
  Change at Day 21: Retardation | -0.63 (3.077) | 0 (1.803)
  Baseline: Said he/she was no good | 0.26 (0.452) | 0.22 (0.441)
  Change at Day 21: Said he/she was no good | 0.05 (0.621) | 0.22 (0.441)
  Baseline: Social competence | 17.37 (3.847) | 17.44 (2.242)
  Change at Day 21: Social competence | 0.11 (2.233) | 0.67 (3.354)
  Baseline: Social interest | 6.84 (3.516) | 8.89 (2.522)
  Change at Day 21: Social interest | 1.16 (3.775) | 1.78 (5.674)
Statistical Analysis 1: Comparison: PF-02545920 15 Milligram (mg) vs Placebo; Change at Day 21: Cried; Test type: Superiority or Other; Median Difference (Net) = -0.158, 90% CI 2-sided [-1.546 to 1.231], Standard Deviation 0.844
Statistical Analysis 2: Comparison: PF-02545920 15 Milligram (mg) vs Placebo; Change at Day 21: Felt blue or depressed; Test type: Superiority or Other; Mean Difference (Net) = 0.444, 90% CI 2-sided [-1.329 to 2.218], Standard Deviation 1.078
Statistical Analysis 3: Comparison: PF-02545920 15 Milligram (mg) vs Placebo; Change at Day 21: Irritability; Test type: Superiority or Other; Mean Difference (Net) = 1.544, 90% CI 2-sided [-5.561 to 8.649], Standard Deviation 4.320
Statistical Analysis 4: Comparison: PF-02545920 15 Milligram (mg) vs Placebo; Change at Day 21: Manifest psychosis; Test type: Superiority or Other; Mean Difference (Net) = 0.573, 90% CI 2-sided [-4.287 to 5.433], Standard Deviation 2.955
Statistical Analysis 5: Comparison: PF-02545920 15 Milligram (mg) vs Placebo; Change at Day 21: Personal neatness; Test type: Superiority or Other; Mean Difference (Net) = 0.556, 90% CI 2-sided [-2.892 to 4.003], Standard Deviation 2.096
Statistical Analysis 6: Comparison: PF-02545920 15 Milligram (mg) vs Placebo; Change at Day 21: Refused to speak; Test type: Superiority or Other; Mean Difference (Net) = -0.327, 90% CI 2-sided [-1.202 to 0.547], Standard Deviation 0.532
Statistical Analysis 7: Comparison: PF-02545920 15 Milligram (mg) vs Placebo; Change at Day 21: Retardation; Test type: Superiority or Other; Mean Difference (Net) = -0.632, 90% CI 2-sided [-5.152 to 3.889], Standard Deviation 2.749
Statistical Analysis 8: Comparison: PF-02545920 15 Milligram (mg) vs Placebo; Change at Day 21: Said he/she was no good; Test type: Superiority or Other; Mean Difference (Net) = -0.170, 90% CI 2-sided [-1.110 to 0.771], Standard Deviation 0.572
Statistical Analysis 9: Comparison: PF-02545920 15 Milligram (mg) vs Placebo; Change at Day 21: Social competence; Test type: Superiority or Other; Mean Difference (Net) = -0.561, 90% CI 2-sided [-4.887 to 3.764], Standard Deviation 2.630
Statistical Analysis 10: Comparison: PF-02545920 15 Milligram (mg) vs Placebo; Change at Day 21: Social interest; Test type: Superiority or Other; Mean Difference (Net) = -0.620, 90% CI 2-sided [-7.934 to 6.694], Standard Deviation 4.447

14. Secondary Outcome: Change From Baseline in Global Assessment of Functioning (GAF) Score at Day 21
Description: GAF is a single clinician-rated item to measure the severity of illness-related impairment in psychological, social and occupational functioning. It is a 100 point rating scale, score range: 0= worst functioning to 99= superior functioning, where higher scores indicates better functioning.
Time Frame: Baseline (Day 1), Day 21
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-02545920 15 Milligram (mg) | Placebo
Number analyzed (Participants) | 22 | 9
units on a scale
  Baseline | 41.18 (10.285) | 40.78 (9.497)
  Change at Day 21 | 8.05 (12.786) | 2.33 (10.677)
Statistical Analysis 1: Comparison: PF-02545920 15 Milligram (mg) vs Placebo; Test type: Superiority or Other; Mean Difference (Net) = 5.712, 90% CI 2-sided [-14.42 to 25.845], Standard Deviation 12.240

15. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 10 days after last dose that were absent before treatment or that worsened relative to pretreatment state. AEs included both serious and non-serious adverse events.
Time Frame: Baseline (Day 1) up to Day 31
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-02545920 15 Milligram (mg) | Placebo
Number analyzed (Participants) | 24 | 11
participants
  Adverse event | 22 | 9
  Serious adverse event | 5 | 0

16. Other Pre Specified Outcome: Number of Participants With Vital Signs of Potential Clinical Concern
Description: Criteria for vital signs of potential clinical concern: pulse rate (supine/sitting position) less than (<) 40 or greater than (>) 120 beats per minute (bpm), pulse rate in standing position <40 or >140 bpm; systolic blood pressure (SBP) <90 millimeters of mercury (mm Hg) and greater than or equal to (>=) 30 mm Hg change (increase, decrease) from baseline in same posture; diastolic blood pressure (DBP) <50 mm Hg and >=20 mm Hg change (increase, decrease) from baseline in same posture.
Time Frame: Baseline (Day 1) up to Day 31
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-02545920 15 Milligram (mg) | Placebo
Number analyzed (Participants) | 24 | 11
participants
  Supine pulse rate <40 bpm | 0 | 0
  Supine pulse rate >120 bpm | 0 | 0
  Standing pulse rate <40 bpm | 0 | 0
  Standing pulse rate >140 bpm | 3 | 2
  Supine SBP <90 mm Hg | 0 | 0
  Standing SBP <90 mm Hg | 1 | 0
  Increase from baseline in supine SBP >=30 mm Hg | 0 | 0
  Increase from baseline in standing SBP >=30 mm Hg | 1 | 0
  Decrease from baseline in supine SBP >=30 mm Hg | 3 | 3
  Decrease from baseline in standing SBP >=30 mm Hg | 2 | 1
  Supine DBP <50 mm Hg | 1 | 0
  Standing DBP <50 mm Hg | 1 | 0
  Increase from baseline in supine DBP >=20 mm Hg | 2 | 0
  Increase from baseline in standing DBP >=20 mm Hg | 4 | 0
  Decrease from baseline in supine DBP >=20 mm Hg | 8 | 2
  Decrease from baseline in standing DBP >=20 mm Hg | 4 | 6

17. Other Pre Specified Outcome: Number of Participants With Clinically Significant Physical and Neurological Examination Abnormalities
Description: Analysis include general physical examination and assessment of head, ears, eyes, ocular fundi, nose, mouth, throat, neck, thyroid, lungs, heart, breasts, abdomen and musculoskeletal and neurological systems. Clinical significance was based on the investigator's discretion.
Time Frame: Baseline (Day 1) up to Day 31
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-02545920 15 Milligram (mg) | Placebo
Number analyzed (Participants) | 24 | 11
participants
  Physical examination | 0 | 0
  Neurological examination | 0 | 0

18. Other Pre Specified Outcome: Number of Participants With Electrocardiogram (ECG) Values of Potential Clinical Concern
Description: Criteria for ECG values for potential clinical concern: PR interval >=300 millisecond (msec), >=25 percent increase when baseline >200 msec, and >=50 percent increase when baseline less than or equal to (<=) 200 msec; QRS interval >=200 msec, >=25 percent increase when baseline >100 msec, and >=50 percent increase when baseline <=100 msec; QTcB interval (corrected QT interval using Bazett's formula) >=500 msec.
Time Frame: Baseline (Day 1) up to Day 31
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-02545920 15 Milligram (mg) | Placebo
Number analyzed (Participants) | 24 | 11
participants | 0 | 0

19. Other Pre Specified Outcome: Number of Participants With Laboratory Abnormalities
Description: Criteria for laboratory abnormalities: Hemoglobin (Hgb), hematocrit, red blood cell (RBC) count: <0.8*lower limit of normal (LLN), platelet: <0.5*LLN or >1.75*upper limit of normal (ULN), white blood cell (WBC): <0.6*LLN or >1.5*ULN, lymphocyte, neutrophil: <0.8*LLN or >1.2*ULN, basophil, eosinophil, monocyte: >1.2*ULN; total bilirubin >1.5*ULN, aspartate aminotransferase, alanine aminotransferase, gamma-glutamyl transferase, alkaline phosphatase: > 3.0*ULN, total protein, albumin: <0.8*LLN or>1.2*ULN; blood urea nitrogen, creatinine: >1.3*ULN, uric acid >1.2*ULN; cholesterol (HDL <0.8*LLN, LDL >1.2*ULN); sodium <0.95*LLN or >1.05*ULN, potassium, chloride, calcium, magnesium, bicarbonate: <0.9*LLN or >1.1*ULN, phosphate <0.8*LLN or >1.2*ULN; prolactin >1.1*ULN; glucose <0.6*LLN or >1.5*ULN, glycosylated hemoglobin >1.3*ULN, creatine kinase >2.0*ULN; urine (pH <4.5 or >8, glucose, ketone, protein, blood/Hgb >=1, RBC, WBC >=6).
Time Frame: Baseline (Day 1) up to Day 31
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-02545920 15 Milligram (mg) | Placebo
Number analyzed (Participants) | 24 | 10
participants | 18 | 8

20. Other Pre Specified Outcome: Number of Participants With Abnormal Prolactin Level
Description: Number of participants with abnormal values (>1.1* ULN) of prolactin level were reported.
Time Frame: Baseline (Day 1) up to Day 21
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-02545920 15 Milligram (mg) | Placebo
Number analyzed (Participants) | 22 | 9
participants | 2 | 0

21. Other Pre Specified Outcome: Number of Participants With Abnormal High Density Lipoprotein (HDL) and Low Density Lipoprotein (LDL) Level
Description: Number of participants with abnormal values of HDL level <0.8* LLN and LDL level >1.2*ULN were reported.
Time Frame: Baseline up to Day 21
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-02545920 15 Milligram (mg) | Placebo
Number analyzed (Participants) | 24 | 10
participants
  HDL <0.8*LLN: number analyzed (Participants) | 22 | 9
  HDL <0.8*LLN | 0 | 1
  LDL >1.2*ULN: number analyzed (Participants) | 21 | 8
  LDL >1.2*ULN | 3 | 0

22. Other Pre Specified Outcome: Number of Participants With Abnormal Glycosylated Hemoglobin (HbA1c) Level
Description: Number of participants with abnormal values (>1.3* ULN) of HbA1c level were reported.
Time Frame: Baseline (Day 1) up to Day 21
Population: Safety analysis set included all participants who received at least 1 dose of study medication. Here, 'N' signifies those participants who were evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | PF-02545920 15 Milligram (mg) | Placebo
Number analyzed (Participants) | 22 | 10
participants | 3 | 0

23. Other Pre Specified Outcome: Number of Participants With Abnormal Fasting Insulin Level
Description: Fasting glucose level below 6 micro international unit per milliliter (mcIU/mL) or above 27 mcIU/mL were considered as abnormal. Number of participants with abnormal values of fasting insulin level were reported.
Time Frame: Baseline (Day 1) up to Day 21
Population: Safety analysis set included all participants who received at least 1 dose of study medication. Here, 'N' signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | PF-02545920 15 Milligram (mg) | Placebo
Number analyzed (Participants) | 24 | 10
participants | 13 | 4

24. Other Pre Specified Outcome: Change From Baseline in Body Weight at Day 21
Time Frame: Baseline (Day 1), Day 21
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: kilogram
Arm/Group | PF-02545920 15 Milligram (mg) | Placebo
Number analyzed (Participants) | 24 | 11
kilogram
  Baseline: number analyzed (Participants) | 23 | 11
  Baseline | 87.48 (28.977) | 85.82 (16.969)
  Change at Day 21: number analyzed (Participants) | 21 | 9
  Change at Day 21 | -1.07 (4.468) | -0.22 (3.567)
Statistical Analysis 1: Comparison: PF-02545920 15 Milligram (mg) vs Placebo; Test type: Superiority or Other; Mean Difference (Net) = -0.849, 90% CI 2-sided [-7.807 to 6.109], Standard Deviation 4.230

25. Other Pre Specified Outcome: Change From Baseline in Abdominal Girth at Day 21
Time Frame: Baseline (Day 1), Day 21
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | PF-02545920 15 Milligram (mg) | Placebo
Number analyzed (Participants) | 24 | 11
centimeter
  Baseline: number analyzed (Participants) | 23 | 11
  Baseline | 86.57 (19.654) | 90.15 (14.87)
  Change at Day 21: number analyzed (Participants) | 21 | 9
  Change at Day 21 | 1.64 (6.701) | 5.83 (13.818)
Statistical Analysis 1: Comparison: PF-02545920 15 Milligram (mg) vs Placebo; Test type: Superiority or Other; Mean Difference (Net) = -4.195, 90% CI 2-sided [-19.50 to 11.114], Standard Deviation 9.307

26. Other Pre Specified Outcome: Change From Baseline in Extrapyramidal Symptom Rating Scale - Abbreviated (ESRS-A) Score at Day 21
Description: ESRS-A is an instrument used to assess extrapyramidal symptoms (including tremor and dystonic reactions). It assesses 4 items: Parkinsonism, dystonia, dyskinesia, and akathisia. Each item is scored on a 5-point severity scale ranging from 0 to 4, with higher score indicating greater severity of symptoms.
Time Frame: Baseline (Day 1), Day 21
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-02545920 15 Milligram (mg) | Placebo
Number analyzed (Participants) | 24 | 11
units on a scale
  Baseline: Parkinsonism: number analyzed (Participants) | 24 | 10
  Baseline: Parkinsonism | 2.5 (2.919) | 1.7 (2.058)
  Change at Day 21: Parkinsonism: number analyzed (Participants) | 11 | 4
  Change at Day 21: Parkinsonism | -0.27 (3.952) | 0 (0.816)
  Baseline: Dyskinesia: number analyzed (Participants) | 24 | 10
  Baseline: Dyskinesia | 0.58 (1.472) | 0.6 (1.075)
  Change at Day 21: Dyskinesia: number analyzed (Participants) | 11 | 4
  Change at Day 21: Dyskinesia | 0.82 (3.371) | 1 (1.155)
  Baseline: Dystonia: number analyzed (Participants) | 24 | 10
  Baseline: Dystonia | 0.29 (1.083) | 0.3 (0.675)
  Change at Day 21: Dystonia: number analyzed (Participants) | 11 | 4
  Change at Day 21: Dystonia | -0.18 (1.401) | 0.75 (1.5)
  Baseline: Akathisia: number analyzed (Participants) | 24 | 10
  Baseline: Akathisia | 0.54 (1.215) | 0.7 (1.337)
  Change at Day 21: Akathisia: number analyzed (Participants) | 11 | 4
  Change at Day 21: Akathisia | 0.45 (1.864) | -0.25 (0.5)
Statistical Analysis 1: Comparison: PF-02545920 15 Milligram (mg) vs Placebo; Change at Day 21: Parkinsonism; Test type: Superiority or Other; Mean Difference (Net) = -0.273, 90% CI 2-sided [-6.010 to 5.465], Standard Deviation 3.488
Statistical Analysis 2: Comparison: PF-02545920 15 Milligram (mg) vs Placebo; Change at Day 21: Dyskinesia; Test type: Superiority or Other; Mean Difference (Net) = -0.182, 90% CI 2-sided [-5.130 to 4.766], Standard Deviation 3.008
Statistical Analysis 3: Comparison: PF-02545920 15 Milligram (mg) vs Placebo; Change at Day 21: Dystonia; Test type: Superiority or Other; Mean Difference (Net) = -0.932, 90% CI 2-sided [-3.275 to 1.411], Standard Deviation 1.425
Statistical Analysis 4: Comparison: PF-02545920 15 Milligram (mg) vs Placebo; Change at Day 21: Akathisia; Test type: Superiority or Other; Mean Difference (Net) = 0.705, 90% CI 2-sided [-2.013 to 3.422], Standard Deviation 1.652

27. Other Pre Specified Outcome: Change From Baseline in Stanford Sleepiness Scale (SSS) Score at Day 4, 7, 14 and 21
Description: SSS is a 7-point Likert scale which facilitates standardized observation of alertness and rates sleepiness, where 1= alert/wide awake, 2= able to concentrate, 3= not at full alertness, 4= not at peak and let down, 5= beginning to lose interest in remaining awake, 6= sleepiness, 7= sleep onset soon; lost struggle to remain awake. Score ranging from 1 to 7, where higher score indicates more sleepiness.
Time Frame: Baseline (Day 1), Day 4, 7, 14, 21
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-02545920 15 Milligram (mg) | Placebo
Number analyzed (Participants) | 24 | 11
units on a scale
  Baseline: number analyzed (Participants) | 23 | 10
  Baseline | 2.3 (0.926) | 2 (1.054)
  Change at Day 4: number analyzed (Participants) | 22 | 10
  Change at Day 4 | -0.09 (1.019) | 0.2 (1.549)
  Change at Day 7: number analyzed (Participants) | 19 | 9
  Change at Day 7 | 0.11 (1.243) | -0.22 (1.563)
  Change at Day 14: number analyzed (Participants) | 13 | 6
  Change at Day 14 | -0.23 (1.536) | -0.67 (1.211)
  Change at Day 21: number analyzed (Participants) | 10 | 4
  Change at Day 21 | -0.4 (1.075) | -0.5 (1.291)
Statistical Analysis 1: Comparison: PF-02545920 15 Milligram (mg) vs Placebo; Change at Day 4; Test type: Superiority or Other; Mean Difference (Net) = -0.291, 90% CI 2-sided [-2.270 to 1.688], Standard Deviation 1.203
Statistical Analysis 2: Comparison: PF-02545920 15 Milligram (mg) vs Placebo; Change at Day 7; Test type: Superiority or Other; Mean Difference (Net) = 0.327, 90% CI 2-sided [-1.892 to 2.547], Standard Deviation 1.349
Statistical Analysis 3: Comparison: PF-02545920 15 Milligram (mg) vs Placebo; Change at Day 14; Test type: Superiority or Other; Mean Difference (Net) = 0.436, 90% CI 2-sided [-1.946 to 2.817], Standard Deviation 1.448
Statistical Analysis 4: Comparison: PF-02545920 15 Milligram (mg) vs Placebo; Change at Day 21; Test type: Superiority or Other; Mean Difference (Net) = 0.100, 90% CI 2-sided [-1.763 to 1.963], Standard Deviation 1.133

28. Other Pre Specified Outcome: Oral Clearance (CL/F) of PF-02545920
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes.
Time Frame: Hour 0 (pre-morning dose) on Day 7, 14, 21; 20 minutes post-dose on Day 7; 1.5, 4.5 hours post-dose on Day 14 and 24 hours post-dose on Day 21
Population: Data was not collected for this outcome measure, due to early termination of the study and the limited number of participants dosed with PF-02545920 resulted in insufficient pharmacokinetic (PK) sampling to support development of a model to calculate the PK parameters.
Arm/Group | PF-02545920 15 Milligram (mg) | Placebo
Number analyzed (Participants) | 0 | 0

29. Other Pre Specified Outcome: Area Under the Concentration Time Curve (AUC) of PF-02545920
Description: AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption.
Time Frame: as for outcome 28
Population: Data was not collected for this outcome measure, due to early termination of the study and the limited number of participants dosed with PF-02545920 resulted in insufficient PK sampling to support development of a model to calculate the PK parameters.
Arm/Group | PF-02545920 15 Milligram (mg) | Placebo
Number analyzed (Participants) | 0 | 0

30. Other Pre Specified Outcome: Steady State Average Concentration of PF-02545920 Over the Dosing Interval (Css,Avg)
Time Frame: as for outcome 28
Population: as for outcome 29
Arm/Group | PF-02545920 15 Milligram (mg) | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | PF-02545920 15 Milligram (mg) | Placebo
Serious Adverse Events (participants affected / at risk) | 5/24 | 0/11
Other Adverse Events (participants affected / at risk) | 22/24 | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-02545920 15 Milligram (mg) (N=24) | Placebo (N=11)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0
Dystonia (Nervous system disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0
Schizophrenia (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | PF-02545920 15 Milligram (mg) (N=24) | Placebo (N=11)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 2
Lip dry (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1
Fatigue (General disorders) | 1 | 0
Influenza like illness (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Tinea pedis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood pressure orthostatic (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 1
Weight decreased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Trismus (Musculoskeletal and connective tissue disorders) | 2 | 0
Akathisia (Nervous system disorders) | 2 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0
Cogwheel rigidity (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Dyskinesia (Nervous system disorders) | 1 | 0
Dystonia (Nervous system disorders) | 9 | 1
Headache (Nervous system disorders) | 6 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Parkinsonism (Nervous system disorders) | 2 | 0
Sedation (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 4 | 2
Syncope (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 1 | 0
Depressive symptom (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 3 | 1
Psychotic disorder (Psychiatric disorders) | 2 | 1
Restlessness (Psychiatric disorders) | 2 | 1
Schizophrenia (Psychiatric disorders) | 1 | 0
Somatic delusion (Psychiatric disorders) | 1 | 0
Epididymal tenderness (Reproductive system and breast disorders) | 1/22 | 0/9 — This event was gender specific.
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Hot flush (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Due to early termination of the study, PK parameters were not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.